CLINICAL TRIAL: NCT05780723
Title: A Randomized Controlled Study of Qinghua Quyu Prescription Rectal Instillation for the Treatment of Ulcerative Colitis
Brief Title: Treatment of Ulcerative Colitis With Rectal Instillation of Qinghua Quyu Prescription(QHQYP)
Acronym: QHQYP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Luqing Zhao, Principal Investigator, Beijing Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Z221100007422094
Record Dates: First submitted 2023-03-08; First posted 2023-03-22 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The TCM group is treated with QHQYP by rectal instillation. (Experimental): QHQYP is decocted in water, with a dose of 100ml each time, and rectal instillation before going to bed, once a night, for 8 weeks.
  Interventions: Drug: Treatment group: Rectal instillation of QHQYP
- The control group is treated with mesalazine enema. (Active Comparator): Mesalazine enema, 4g/tube, 1 tube each time, enema before bed, once a night, for 8 weeks.
  Interventions: Drug: Control group: Mesalazine enema treatment

INTERVENTIONS:
Drug: Treatment group: Rectal instillation of QHQYP — QHQYP is decocted in water, with a dose of 100ml each time, and rectal drip before going to bed, once a night, for 8 weeks.
  Other Names: QHQYP is prepared by unified decocting from the Pharmacy Department of Beijing Hospital of Traditional Chinese Medicine, Capital Medical University.
  Arms: The TCM group is treated with QHQYP by rectal instillation.
Drug: Control group: Mesalazine enema treatment — Mesalazine enema, 4g/tube, 1 tube each time, enema before bed, once a night, a total of 8 weeks of continuous treatment.
  Other Names: Mesalazine enema is produced by Vifor AG Zweigniederlassung Medichemie Ettingen, National medicine approval H20150127.
  Arms: The control group is treated with mesalazine enema.

SUMMARY:
This study will enroll 60 patients with mild to moderate active ulcerative colitis as subjects. They will be randomly divided into two groups: the TCM group received QHQYP rectal instillation, while the control group received mesalazine enema. The treatment period for both groups was 8 weeks. The modified Mayo Activity Index will be used as the main evaluation index. Secondary evaluation indices will include the Underwater Endoscopic Severity Index (UCEIS) score, endoscopic Baron score, mucosal histological score (Geboes index), Chinese medicine syndrome efficacy evaluation, quality of life score, physicochemical indicators reflecting disease activity or remission, intestinal microbiota indicators, and changes in inflammation and immune-related indicators in colonoscopy biopsy tissues. Safety indicators were also monitored.

ELIGIBILITY:
Inclusion Criteria:

1. Meets the diagnostic criteria for active ulcerative colitis, with clinical severity being mild or moderate and the lesion range being limited to the rectum or left colon and not extending beyond the splenic flexure.
2. Traditional Chinese medicine diagnosis indicates the presence of damp-heat syndrome in the large intestine.
3. Between the ages of 18 and 65, regardless of gender.
4. Informed consent and voluntary participation are required. The process of obtaining informed consent should comply with GCP regulations.

Exclusion Criteria:

1. Patients with severe disease condition.
2. Patients with infectious colonic diseases such as chronic schistosomiasis, bacterial dysentery, amoebic dysentery, intestinal tuberculosis, as well as non-infectious colonic diseases such as Crohn's disease, ischemic bowel disease, and radiation enteritis.
3. Patients with serious complications such as local stenosis, intestinal obstruction, intestinal perforation, rectal polyps, toxic megacolon, colon cancer, rectal cancer, and anal diseases.
4. Pregnant or lactating women.
5. Patients with severe primary heart, liver, lung, kidney, blood or other severe diseases that affect their survival.
6. Patients with disabilities as defined by law (blind, deaf, mute, intellectually disabled, mentally ill, physically disabled).
7. Patients with suspected or confirmed history of alcohol or drug abuse.
8. Other conditions that may reduce the likelihood of enrollment or complicate enrollment, as determined by the researcher, such as frequent changes in work environment that may lead to loss of follow-up.
9. Patients with allergies to two or more drugs or foods, or with a history of allergy to the components of this medication.
10. Patients currently participating in other clinical trials of medications.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-04-04 (Actual); Primary Completion 2024-10-23 (Actual); Study Completion 2024-10-23 (Actual)

PRIMARY OUTCOMES:
Change from Modified Mayo Activity Index at 8 weeks of treatment | Evaluation will be made at baseline and 8 weeks of treatment.
  To understand the remission status of ulcerative colitis from the stool frequency, rectal bleeding, colonic mucosa condition and physician's overall evaluation. Each of the above aspects includes four levels (from 0 to 3, with higher scores indicating more severe disease).

SECONDARY OUTCOMES:
Change from Ulcerative Colitis Endoscopic Index of Severity(UCEIS) at 8 weeks of treatment | Evaluation will be made at baseline and 8 weeks of treatment.
  It focuses on three aspects: vascular pattern, bleeding and erosions&ulcers. The total score of the three scores can range from 0-8 (normal: 0, mild activity: 1-3, moderate activity: 4-6, and severe activity: 7-8.
Change from Endoscopic Baron score at 8 weeks of treatment | Evaluation will be made at baseline and 8 weeks of treatment.
  To understand the degree of activity of endoscopic ulcerative colitis.It includes four levels (from 0 to 3, with higher scores indicating more severe disease).
Change from Geboes Score at 8 weeks of treatment | Evaluation will be made at baseline and 8 weeks of treatment.
  To understand the status of mucosal tissue score. It ranges from Grade 0 (Architectural changes) , Grade 1 (chronic inflammatory cell infiltration), Grade 2 (neutrophils and eosinophils), Grade 3 (epithelial neutrophils) , Grade 4 (crypt destruction) to Grade 5 (erosion and ulcer). The higher the Geboes score, the more serious the disease activity. A grade lower than 2A.0 can be regarded as histological remission.
Change from Evaluation of curative effect of traditional Chinese medicine syndrome at 8 weeks of treatment | Evaluation will be made at baseline and 2,4,8 weeks of treatment.
  Traditional Chinese medicine (TCM) syndrome score of ulcerative colitis will be carried out to understand whether the symptoms of patients improved after treatment. It consists of 9 questions, and the total scores are ranging from 0 to 43 with higher scores indicating more severe disease.
Change from Quality of life score at 8 weeks of treatment | Evaluation will be made at baseline and 8 weeks of treatment.
  To understand the quality of life score of patients. It consists of 32 questions divided into four dimensions: bowel symptoms (10 items), systemic symptoms (5 items), emotional function (12 items) and social function (5 items). Every question has graded responses from 1 (worst situation) to 7 (best situation), and thus the total score is ranging from 32 to 224 with higher scores representing better quality of life.
Change from Intestinal flora at 8 weeks of treatment | Examination will be performed at baseline and 8 weeks of treatment.
  Fresh feces are collected at baseline and 8 weeks of treatment, and the distribution of intestinal flora is detected by 16s rRNA sequencing technology.

OTHER OUTCOMES:
Change from Inflammation and immune-related indicators in colonoscopy biopsy tissues at 8 weeks of treatment | Examination will be performed at baseline and 8 weeks of treatment.
  Colonoscopy biopsy tissues are collected at baseline and 8 weeks of treatment, and the Inflammation and immune-related indicators is detected by immumohistochemical staining.

CONTACTS AND LOCATIONS:
Overall Officials: Luqing Zhao, Doctor, Principal Investigator — Beijing Hospital of Traditional Chinese Medicine
Locations (1):
- Beijing Hospital of Traditional Chinese Medicine, Capital Medical University, Dongcheng, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ng SC, Shi HY, Hamidi N, Underwood FE, Tang W, Benchimol EI, Panaccione R, Ghosh S, Wu JCY, Chan FKL, Sung JJY, Kaplan GG. Worldwide incidence and prevalence of inflammatory bowel disease in the 21st century: a systematic review of population-based studies. Lancet. 2017 Dec 23;390(10114):2769-2778. doi: 10.1016/S0140-6736(17)32448-0. Epub 2017 Oct 16. PMID 29050646
- [Background] Jones GR, Lyons M, Plevris N, Jenkinson PW, Bisset C, Burgess C, Din S, Fulforth J, Henderson P, Ho GT, Kirkwood K, Noble C, Shand AG, Wilson DC, Arnott ID, Lees CW. IBD prevalence in Lothian, Scotland, derived by capture-recapture methodology. Gut. 2019 Nov;68(11):1953-1960. doi: 10.1136/gutjnl-2019-318936. Epub 2019 Jul 11. PMID 31300515
- [Background] Ahmad R, Sorrell MF, Batra SK, Dhawan P, Singh AB. Gut permeability and mucosal inflammation: bad, good or context dependent. Mucosal Immunol. 2017 Mar;10(2):307-317. doi: 10.1038/mi.2016.128. Epub 2017 Jan 25. PMID 28120842
- [Background] Wu Y, Tang L, Wang B, Sun Q, Zhao P, Li W. The role of autophagy in maintaining intestinal mucosal barrier. J Cell Physiol. 2019 Nov;234(11):19406-19419. doi: 10.1002/jcp.28722. Epub 2019 Apr 24. PMID 31020664
- [Background] Li Q, Cui Y, Xu B, Wang Y, Lv F, Li Z, Li H, Chen X, Peng X, Chen Y, Wu E, Qu D, Jian Y, Si H. Main active components of Jiawei Gegen Qinlian decoction protects against ulcerative colitis under different dietary environments in a gut microbiota-dependent manner. Pharmacol Res. 2021 Aug;170:105694. doi: 10.1016/j.phrs.2021.105694. Epub 2021 Jun 2. PMID 34087350